CLINICAL TRIAL: NCT05807919
Title: Evaluate and Compare the Clinical Efficacy of the Mediterranean Diet to the Low-FODMAP Diet in Treating Irritable Bowel Syndrome
Brief Title: Evaluating the Efficacy of the Mediterranean Diet to the Low- Fermentable, Oligosaccharides, Disaccharides, Monosaccharides, and Polyols (FODMAP) Diet in Treating Irritable Bowel Syndrome(IBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: ModifyHealth (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Prashant Singh, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00227491; 5P30DK089503-13 (NIH)
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Low FODMAP Diet; Mediterranean Diet
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Subjects meeting all eligibility criteria will be randomized in a 1:1 ratio to receive either the MD or the LFD for a four-week period.
Who Masked: Participant, Investigator
Masking Description: Participant and investigators will not know what study cohort participants have been randomized into.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet low in all FODMAP groups (Experimental)
  Interventions: Other: Diet low in all FODMAP groups
- Diet - Mediterranean (Experimental)
  Interventions: Other: Diet - Mediterranean

INTERVENTIONS:
Other: Diet low in all FODMAP groups — Randomized participants will eat this diet for 4 weeks (all meals and snacks will be provided). Participants will only eat the study food for this intervention. Participants will be asked to complete surveys, food diaries, and have blood and stools samples pre and post treatment.
  Arms: Diet low in all FODMAP groups
Other: Diet - Mediterranean — Randomized participants will eat this diet for 4 weeks (all meals and snacks will be provided). Participants will only eat the study food for this intervention. Participants will be asked to complete surveys, food diaries, and have blood and stools samples pre and post treatment.
  Arms: Diet - Mediterranean

SUMMARY:
This study is being completed to determine if the Mediterranean (MD) and low FODMAP (fermentable, oligosaccharides, disaccharides, monosaccharides, and polyols) diets are comparable in the effectiveness to treat Irritable Bowel Syndrome (IBS).

The study team hypothesizes that:

* The low FODMAP and Mediterranean groups will achieve a similar improvement in abdominal pain
* Both groups will achieve similar improvements in bloating, overall IBS symptom severity, and adequate relief

ELIGIBILITY:
Inclusion Criteria:

* Patients with IBS-D (diarrhea-predominant IBS) or IBS-M (IBS with mixed subtype) diagnosed per Rome IV questionnaire and without any unexplained alarm features (rectal bleeding, weight loss, nocturnal symptoms, personal history of celiac disease, microscopic colitis, inflammatory bowel disease)
* Aged 18-70 years at the time of screening
* Weekly average of worst daily (in the past 24 hours) abdominal pain score of ≥3.0 on a 0-to-10-point scale
* At least 80 percent compliance in daily questionnaire entries during the 7-day screening period

Exclusion Criteria:

* Subjects adhering to any dietary IBS treatment such as the low-fodmap diet, or gluten-free diet, Mediterranean currently or within the past 6 months
* Subjects with a known food allergy to eggs, seafood, peanuts, tree nuts or milk (subjects with lactose intolerance that are experiencing IBS symptoms while on a lactose-free diet will not be excluded from the study).
* Subjects with a history of poorly controlled insulin-dependent or non-insulin-dependent diabetes
* Subjects with a known history of organic Gastrointestinal (GI) disease (i.e., celiac disease, inflammatory bowel disease or microscopic colitis)
* Subjects with a history of an eating disorder requiring medical or behavioral treatment within the past 10 years.
* Subjects with prior small bowel or colonic surgery (excluding appendectomy or cholecystectomy if over 6 months since these 2 procedures)
* Oral antibiotic use in the past 3 months
* Any planned significant changes in dietary or exercise regimen within 30 days prior to Screening or during the study.
* Currently pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Singh, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh P, Dean G, Iram S, Peng W, Chey SW, Rifkin S, Lothen-Kline C, Muir J, Lee AA, Eswaran S, Chey WD. Efficacy of Mediterranean Diet vs. Low-FODMAP Diet in Patients With Nonconstipated Irritable Bowel Syndrome: A Pilot Randomized Controlled Trial. Neurogastroenterol Motil. 2025 Oct;37(10):e70060. doi: 10.1111/nmo.70060. Epub 2025 Apr 24. PMID 40273380

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diet Low in All FODMAP Groups | Diet - Mediterranean
Started | 11 | 15
Actual Treatment Begun (Day 1) | 11 | 14
Elected to Continue Treatment After Day 1 | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 5
Not completed — Received antibiotics - excluded | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Ethnicity data was not collected for this trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Diet Low in All FODMAP Groups | Diet - Mediterranean | Total
Number analyzed (Participants) | 11 | 15 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.09 (19.5) | 38.13 (11.3) | 41.1 (15.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 1 | 1 | 2
  Non-Binary | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 11 | 15 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 10 | 11 | 21
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Are Responders Based on the Abdominal Pain Intensity Score for at Least 2 of 4 Weeks
Description: Results reflect the participants who were weekly responders for at least 2 of the 4 weeks based on their abdominal pain intensity score. The abdominal pain score was a single-question, 11-point numeric rating scale in which 0 represented no abdominal pain and 11 represented the worst possible abdominal pain. Once per day, subjects reported their worst daily (in the past 24 hours) abdominal pain. A weekly responder was defined as a participant whose score decreased in the weekly average of worst abdominal pain in the past 24 hours by at least 30% compared with baseline.
Time Frame: 4 weeks
Population: Results are based on a modified intent to treat (mITT) analysis. Participants categorized in the Participant Flow as "Withdrawal by Subject" were not included in the mITT analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Diet Low in All FODMAP Groups | Diet - Mediterranean
Number analyzed (Participants) | 11 | 11
Participants | 9 | 8
Statistical Analysis 1: Comparison: Diet Low in All FODMAP Groups vs Diet - Mediterranean; Test type: Superiority; p = 1.00, Fisher Exact

2. Secondary Outcome: Proportion of Participants Who Are Weekly Responders to Adequate Relief Symptom Assessment for at Least 2 of 4 Weeks
Description: Results reflect the participants who were weekly responders based on the adequate relief symptom assessment for at least 2 of the 4 weeks. Participants provided a binary (yes or no) response to rate the adequacy of relief of global irritable bowel syndrome (IBS) symptoms at the start of the study and weekly thereafter. A weekly responder was defined as a participant who achieved adequate relief in symptoms in at least 2 out of 4 weeks of the treatment period.
Time Frame: 4 weeks
Population: Results are based on a mITT analysis. Participants categorized in the Participant Flow as "Withdrawal by Subject" were not included in the mITT analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Diet Low in All FODMAP Groups | Diet - Mediterranean
Number analyzed (Participants) | 11 | 11
Participants | 6 | 3
Statistical Analysis 1: Comparison: Diet Low in All FODMAP Groups vs Diet - Mediterranean; Test type: Superiority; p = 0.39, Fisher Exact

3. Secondary Outcome: Proportion of Participants Who Are Weekly Responders Based on the Irritable Bowel Severity Scoring System (IBS-SSS) Modified Version for at Least 2 of the 4 Weeks
Description: Results reflect participants who were weekly responders for at least 2 of the 4 weeks based on their scores on a modified version of the IBS-SSS. This version of the IBS-SSS was comprised of 5 questions participants answered based on their stomach and bowels. The total score for this modified version of the IBS-SSS was 0-500, with 0 indicating no IBS symptoms and 500 indicating the highest amount of IBS symptoms. A weekly responder was defined as a participant whose score decreased in the weekly IBS-SSS by at least 50 points compared with baseline.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Diet Low in All FODMAP Groups | Diet - Mediterranean
Number analyzed (Participants) | 11 | 11
Participants | 9 | 5
Statistical Analysis 1: Comparison: Diet Low in All FODMAP Groups vs Diet - Mediterranean; Test type: Superiority; p = 0.18, Fisher Exact

4. Secondary Outcome: Change in Mean Score of the Irritable Bowel Severity Scoring System (IBS-SSS) Modified Version
Description: The modified version of the IBS-SSS was comprised of 5 questions participants answered based on their stomach and bowels. The total score for this modified version of the IBS-SSS was 0-500, with 0 indicating no IBS symptoms and 500 indicating the highest amount of IBS symptoms. The results represent the mean change from baseline minus 4 weeks.
Time Frame: Baseline, 4 weeks
Population: Results are based on a per-protocol analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Diet Low in All FODMAP Groups | Diet - Mediterranean
Number analyzed (Participants) | 10 | 10
score on a scale | -105.5 [-260 to -66] | -60 [-227 to 57]
Statistical Analysis 1: Comparison: Diet Low in All FODMAP Groups vs Diet - Mediterranean; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Proportion of Participants Who Are Weekly Responders to Bloating for at Least 2 of the 4 Weeks
Description: Results reflect the number of participants who were weekly responders based on their abdominal bloating score for at least 2 of 4 weeks. The abdominal bloating score was a single-question, 11-point numeric rating scale in which 0 represented no abdominal bloating and 11 represented the worst possible abdominal bloating. Once per day, participants reported their worst daily (in the past 24 hours) abdominal bloating. A weekly responder was defined as a participant whose score decreased in the weekly average of worst bloating in the past 24 hours by at least 30% compared with baseline.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Diet Low in All FODMAP Groups | Diet - Mediterranean
Number analyzed (Participants) | 11 | 11
Participants | 8 | 5
Statistical Analysis 1: Comparison: Diet Low in All FODMAP Groups vs Diet - Mediterranean; Test type: Superiority; p = 0.39, Fisher Exact

6. Secondary Outcome: Participants Who Are Weekly Responders to Stool Consistency Based on the Bristol Stool Scale (BSS) for at Least 2 of the 4 Weeks
Description: Results reflect the participants who were weekly responders based on their stool consistency assessment for at least 2 of 4 weeks. A stool consistency weekly responder was defined as a participant with a 50% or greater reduction in the number of days per week with at least one abnormal stool. Stools that scored as 1 or 2 (hard stool) or 6 or 7 (liquid stool) on the BSS were defined as abnormal.
Time Frame: 4 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Diet Low in All FODMAP Groups | Diet - Mediterranean
Number analyzed (Participants) | 11 | 11
Participants | 2 | 0
Statistical Analysis 1: Comparison: Diet Low in All FODMAP Groups vs Diet - Mediterranean; Test type: Superiority; p = 0.48, Fisher Exact

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Diet Low in All FODMAP Groups | Diet - Mediterranean
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15
Other Adverse Events (participants affected / at risk) | 1/11 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diet Low in All FODMAP Groups (N=11) | Diet - Mediterranean (N=15)
Worsening Constipation (Gastrointestinal disorders) | 1 | 0
Worsening Abdominal Pain (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT05807919/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT05807919/ICF_001.pdf